CLINICAL TRIAL: NCT06794307
Title: Blood Glucose Levels in Pregnant Non-diabetic Women During Treatment With Betamethasone for Fetal Lung Maturation
Brief Title: Blood Glucose in Pregnant Non-diabetic Women During Treatment With Betamethasone for Fetal Lung Maturation
Status: Recruiting | Type: Observational
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Other Study IDs: 2024_VB_CGM
Record Dates: First submitted 2024-10-21; First posted 2025-01-27 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Preterm Birth; Hyperglycemia; Neonatal Hypoglycemia; Threatened Preterm Labor
Keywords: Preterm birth; Betamethasone; Continuous glucose monitoring; Antenatal corticosteroids
MeSH Terms: conditions — Premature Birth; Hyperglycemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples Without DNA — serum, plasma, umbilical cord blood, urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
In case of threatening preterm birth, it is standard to recommend treatment with betamethasone to accelerate fetal lung maturation. In pregnant women with diabetes, treatment with betamethasone can lead to significant hyperglycemia, which may cause hypoglycemia in the neonate. Changes in blood glucose in non-diabetic women are less investigated. In this study we aim to examine changes in maternal blood glucose levels in non-diabetic women, during treatment with betamethasone, by continuous glucose monitoring.

Hypotheses:

Administration of betamethasone induce significant hyperglycemia in non-diabetic pregnant women during treatment.

DETAILED DESCRIPTION:
Antenatal corticosteroid administration is an important treatment to reduce the incidence of neonatal respiratory distress syndrome, and improve neonatal outcomes of babies born premature.

Administration of betamethasone however also affects the maternal glucose homeostasis, and it is well-known that in pregnant women with diabetes, the administration of glucocorticoids can lead to significant maternal hyperglycemia, and hypoglycemia in the neonate, unless the insulin dosage is adjusted accordingly. Administration of betamethasone also affects the glucose homeostasis in pregnant non-diabetic women. However, only few studies have investigated the changes in the blood glucose levels in non-diabetic pregnant women, and a more accurate depiction of the glycemic response to betamethasone can be obtained by continuous glucose monitoring.

Recruitment of participants will occur upon their arrival with symptoms of threatened preterm birth, when it is decided to start treatment with betamethasone for fetal lung maturation.

To measure blood glucose levels in the pregnant women, a continuous glucose monitor (CGM) will be used.

Further, blood samples will be collected on days 1-6 after inclusion, for measurement of: Insulin, blood glucose, 3-hydroxybutyrat, HgbA1c, CRP and leucocytes.

Urine dipstick test for ketones and glucose will be performed twice daily. After delivery, a blood sample will be extracted from the umbilical cord for measurement of Ph, base-excess, glucose, insulin c-peptide and inflammatory markers.

Information on hypoglycemia and/or the need for early feeding of the infant after birth will be recorded.

Perspectives:

The results of this study will help us understand how the administration of betamethasone affects maternal blood glucose levels. If it is found, that administration of betamethasone causes significant hyperglycemia in the pregnant women, it may be important to measure and treat hyperglycemia during betamethasone treatment, to ensure the effect of betamethasone and prevent neonatal complications due to hypoglycemia.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant in gestational week 24+0 - 34+0 admitted with symptoms of threatened preterm birth:

  * Premature contractions and shortening of the cervix, or
  * Preterm premature rupture of membranes.
* Treatment with betamethasone for fetal lung maturation is planned, or started (maximum 4 hours before inclusion)
* Age over 18 years
* Read and understand Danish

Exclusion Criteria:

* Multiple pregnancy
* Diabetes
* Pre-existing maternal use of medications that affect glucose metabolism

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Pregnant women
Study Population: Pregnant women admitted with symptoms of threatened preterm birth in gestational week 24+0 - 34+0
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2024-11-20 (Actual); Primary Completion 2025-10-30 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Maternal blood glucose levels before, under and after the administration of betamethasone | 7-14 days
  Blood glucose levels (mmol/L) will be measured continuously using a continuous glucose monitor including a small electrode under the skin

SECONDARY OUTCOMES:
The level of insulin (pmol/L)in maternal blood before, during, and after the effect of betamethasone | 7 days. From the day betamethasone is given untill 6 days after the first dose
  Blood samples will be collected on days 1-6, where day 1 is the day where the first dose of betamethasone is given.
The level of 3-hydroxybuturat (mmol/L) in maternal blood before, during and after treatment with Betamethasone | 7 days. From the day betamethasone is given untill 6 days after the first dose
  Blood samples will be collected on days 1-6, where day 1 is the day where the first dose of betamethasone is given.
Level of leukocytes (White blood cell count) (mia/L) in maternal blood before, during and after treatment with betamethasone | 7 days, from day one (the day where the first dose of betamethasone is given) untill 6 days after the first dose.
  Blood samples will be collected on days 1-6, where day 1 is the day where the first dose of betamethasone is given.
The level of CRP (C-reactive protein)(nmol/ml) in maternal blood before, during and after treatment with betamethasone | 7 days. From the day betamethasone is given untill 6 days after the first dose.
  Blood samples will be collected on days 1-6, where day 1 is the day where the first dose of betamethasone is given.
The level of glucose (mmol/L) in umbilical cord blood at delivery | At delivery of the baby
  After the birth and cord occlusion a blood sample will be drawn from the umbilical cord
The level of insulin (pmol/L) in umbilical cord blood at delivery | At delivery
  After the birth and cord occlusion a blood sample will be drawn from the umbilical cord
The level of c-peptid (pmol/L) in umbilical cord blood at delivery | At delivery
  After the birth and cord occlusion a blood sample will be drawn from the umbilical cord
The level af adiponectin (ug/ml) in umbilical cord blood at delivery | At delivery
  After the birth and cord occlusion a blood sample will be drawn from the umbilical cord
The level of leptin (ng/ml) in umbilical cord blood at delivery | At delivery
  After the birth and cord occlusion a blood sample will be drawn from the umbilical cord
Number of infants with need for early feeding (yes/no) after birth | First two days after birth
  Information from files on whether the infant was given "Early feeding" after delivery (yes/no)

CONTACTS AND LOCATIONS:
Locations (1):
- Aarhus University Hospital, Aarhus, Central Region Denmark, Denmark

IPD SHARING:
Plan to Share IPD: No
No plan decided yet